CLINICAL TRIAL: NCT06127511
Title: Peanut Consumption on Cognitive Performance, Weight Management, and Inflammation in Young Adolescents
Brief Title: Peanut Consumption on Cognitive, Weight, and Inflammation
Acronym: PEANUTY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Gasol Foundation (Unknown); Universitat Oberta de Catalunya (Other); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Responsible Party: Principal Investigator, Rosa M Lamuela-Raventós, Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PEANUTY
Record Dates: First submitted 2023-10-31; First posted 2023-11-13 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Performance; Inflammation; Weight Change, Body; Adolescents
Keywords: peanut; cognitive; inflammation; weight; adolescent; obesity; gut microbiota; healthy dietary; physical activity; sleeping; behaviour habits; Mediterranean diet
MeSH Terms: conditions — Inflammation; Body Weight Changes; Body Weight; Obesity; Motor Activity | interventions — Food

STUDY DESIGN:
Intervention Model Description: A multi-school, two-arm parallel cluster-randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peanuty group (Experimental): Families allocated in the intervention group will receive the whole skin roasted peanuts packed in daily doses (25 g per day, 750 g per month), starting the day that we will visit the participants for the first time. They will consume 25 g of whole skin roasted peanuts as a daily snack to be incorporated into their diet for six months.
  Interventions: Other: Food (peanut)
- Control group (No Intervention): Usual care

INTERVENTIONS:
Other: Food (peanut) — After the recruitment, the participants will follow a peanut-free diet for two weeks.
  Arms: Peanuty group

SUMMARY:
A multi-school, two-arm parallel cluster-randomized controlled trial will be conducted in 200 healthy young adolescents from Barcelona (Spain) to evaluate the effect of peanut consumption on cognitive performance, weight management and inflammation. Schools willing to participate will be randomly assigned to either the intervention or the control group. After the recruitment, the participants will follow a peanut-free diet for two weeks. Both arms will receive a multidimensional educational intervention designed by the Gasol Foundation to promote healthy dietary habits based on Mediterranean diet recommendations, along with exercise performance, healthy sleeping habits and emotional knowledge. Half of the participants (intervention group) will consume 25 g of whole skin roasted peanuts as a daily snack to be incorporated into their diet for six months.

DETAILED DESCRIPTION:
Background:

Regular nut consumption has been associated with reduced inflammation, oxidative damage, and improved vascular function, which may benefit cognitive function. Their content in phenolic acids, mainly p-coumaric and isoferulic acids may help prevent and cure diseases including Alzheimer's, diabetes, cancer, hypertension, and atherosclerosis that are associated with oxidative stress suggesting it could be used as a potential new neuroprotective tactic. Polyphenols have been shown to influence gut microbiota composition and activity, and their metabolites, including short-chain fatty acids (SCFAs), may modulate brain biochemistry by acting as neurotransmitters in the central nervous system, potentially leading to effects against depression and neurodegenerative disease.

Childhood is an important period for brain development, and nutrients aid the formation of new synaptic connections and support learning processes at school and in home environments. Adolescence is also a period where brain connectivity and complex behaviours are further refined. While a positive association has been observed between the consumption of healthy foods (fruits, vegetables, whole grains, fish, nuts, dietary fiber) and cognitive function, research on the association between nut consumption and cognitive health during adolescence is scarce.

In addition, evidence shows that incorporating peanut and peanut-based products into the diet does not lead to weight gain or higher body weight and may even promote long-term weight maintenance and increase linear growth due to their arginine content.

Due to the potential benefits of schools in preventing overweight and obesity, and the lack of research on the relationship between nut consumption and cognitive health during childhood and adolescence, the investigators plan to conduct an intervention study to investigate the association between peanut consumption and cognitive ability, weight management and inflammation in Spanish children aged 10-12 years. As the nutritional composition of peanuts can vary depending on their form, this study will examine the impact of the regular consumption of 25g of whole-skin roasted peanuts on cognitive function, mood, and school performance in healthy young adolescents.

Study design:

A multi-school, two-arm parallel cluster-randomized controlled trial will be conducted in 200 healthy young adolescents from Barcelona (Spain) to evaluate the effect of peanut consumption on cognitive performance, weight management and inflammation. Schools willing to participate will be randomly assigned to either the intervention or the control group. After the recruitment, the participants will follow a peanut-free diet for two weeks. Both arms will receive a multidimensional educational intervention designed by the Gasol Foundation to promote healthy dietary habits based on Mediterranean diet recommendations, along with exercise performance, healthy sleeping habits and emotional knowledge. Half of the participants (intervention group) will consume 25 g of whole skin roasted peanuts as a daily snack to be incorporated into their diet for six months.

Sample size:

Our study is designed based on previous research findings that suggest peanut consumption could influence cognitive performance and adiposity. Using a cluster design, the investigators aim to detect a significant difference of 1.3 (SD 0.8) absolute points in body mass per kJ consumed and a 6.9-unit (SD 3.1) improvement in cognitive performance score between the intervention and control groups, at a 95% confidence level, 80% power, and an estimated number of 20-40 students per school. With an intra-class correlation coefficient of 0.02, the investigators estimated a sample size of 6 schools (3 per arm) with a total of 200 participants (100 in each arm) at baseline, allowing for a 10% drop-out rate.

Ethical aspects:

The project will be submitted to the Research Ethics Committees of the Hospital Clinic and from Barcelona University (UB). Parents or guardians of the participants will sign an informed consent prior to the start. The study will be registered at clinicaltrials.gov. Although the recommended diet is based on the Mediterranean Diet and lifestyle intervention are safe, the investigators will be aware of any side effects in all visits to the participants. Regarding data confidentiality, Spanish Personal Data Protection Law (LOPD 15/99) compliance, all questionnaire data and biological samples pertaining to the participants will be anonymized and coded by a unique ID number. Data will be processed confidentially respecting the basic ethical principles of research that involves the usage of biological samples as established by Law 14/2007 on Biomedical Research and according to the Organic Law 15/1999 (concerning Data Protection), Law 41/2002 (concerning Patient Autonomy) and the Law 14/1986.

Recruitment and randomization:

The study will begin by contacting several schools in Barcelona to inform them about the trial. Each school's allocation group will be notified of its status by email. Then, the investigators will provide the schools with a recruitment flier to assess willingness to collaborate and grant us permission to contact interested families. Trained personnel will then contact the parents and explain the study details. Fieldworkers will review each candidate's eligibility criteria to ensure compliance with the study protocol. Participation in the study will be contingent upon obtaining informed consent from both the parents or guardians of the children and the teachers.

Implementation and adherence:

The healthy lifestyle intervention for all participants (intervention and control groups) This intervention had been developed and tried before as part of the SEÍSMO project by the Gasol Foundation. The SEÍSMO project is an intervention addressed to school-age children (6- to 12-year-old), their parents/caregivers, teaching, and non-teaching staff. It is part of a Multilevel Multicomponent intervention aimed to prevent overweight and obesity from early ages, and along all the developmental stages, until adulthood. The intervention includes 2 main modules: physical education module (PEM) and family module (FAM). The PEM includes a pedagogical guide that considers healthy eating, physical and sport, screen time, sleep duration, and phycological wellbeing in movement. The FAM, which is led by tutors, joins the PEM to increase the efficacy of the project because the family role is necessary to change habits. This includes family home activities, tutoring with the children, motivational messages, video tips about healthy habits for families and a healthy closing event. The family home activities combine with the PEM and each of them consists of a healthy habit promotion. The control group will be asked to refrain from eating nuts.

At the beginning of the intervention, all the educators from participant schools will receive a training to empower them toward healthy habits educational actions. After that, the modules of the SEÍSMO project will be deployed within children, families and the whole educative community.

The peanut intervention:

Families allocated in the intervention group will receive the whole skin roasted peanuts packed in daily doses (25 g per day, 750 g per month), starting the day that the investigators will visit the participants for the first time.

Adherence compliance:

Peanuts will be delivered every two months to keep in contact with the families and who will be asked to fill in a compliance form. To increase the success rate, the investigators will offer recipes with peanuts regularly and in different forms, mainly videos and infographics. the investigators will ask parents to supervise the intervention by checking the subject's adherence to peanuts consumption. Participants in the intervention group will be contacted in the middle of the study.

Data collection:

Trained professionals (nurses and nutritionists) will be in charge to collect participant characteristics at baseline and after 6 months (end of study), and will guide the adolescents through the questionnaires, perform measurements, and collect samples during school hours. Assessment of the characteristics will include a detailed assessment of health behaviors and health factors, including the following: anthropometry and body composition; diet; physical activity; emotion management; biochemical measurements. The assessment at the family and school environment levels will include surveys and questionnaires. Families and school principals will complete online questionnaires sent by e-mail or regular mail if necessary.

Assessment of the participant characteristics and outcomes:

* To evaluate the cognitive skills. Participants will be assessed at baseline and after the intervention by several validated cognitive tests and behavioural rating scales. Changes from baseline in the main score for each of the tests for neuropsychological (working memory, attention, fluid intelligence, and executive function) and behavioral outcomes will be measured using a total of 4 tests designed for evaluating children and adolescents: N-back task, the Attention Network Test (ANT), the Tests of Primary Mental Abilities (PMA-R, the Spanish adaptation), the Roulettes Task (adapted from the Cups Task), and the Strengths and Difficulties Questionnaire (SDQ).
* To evaluate the body composition, diet, and clinical status of volunteers. Anthropometric measurements (weight, height, body mass index, waist and hip circumference, body fat %, muscle mass %, visceral fat, fat mass index, lean mass index) will be measured and expressed as z-score by age and sex. Clinical parameters (blood pressure and heart rate) and biochemical analysis (lipid profile and, glucose) in fasting blood will be measured. A 16-item Mediterranean Diet Quality Index Questionnaire for Spanish Adolescents (KIDMED) and an FFQ validated for the Spanish population and adapted to the adolescent population will be used to evaluate the participants' diet. Physical activity and sleep will be measured through validated questionnaires and by accelerometery. Onset and progression of pubertal changes will be measured by Tanner self-assessment questionnaire.
* To evaluate the prebiotic and postbiotic effects, the investigators will collect capillary blood micro-samples, faeces and urine samples. By using these minimally invasive sampling methods, the investigators aim to minimise any discomfort for the participants to determine:

  * Microbial phenolic metabolites in urine samples. A novel and validated targeted metabolomics method based on liquid chromatography coupled to high-resolution mass spectrometry will be used to identify and quantify microbial phenolic metabolites.
  * Short-chain fatty acids in faecal samples. Their quantification will be performed using a headspace sampler connected to a gas chromatography-mass spectrometry system (HS-GC-MS) according to a previously described methodology.
  * Gut microbiota characterization by 16s metagenomic analysis will be performed by experts from the Biomedical Research Institute of Malaga (IBIMA).
* To determine and evaluate the biomarkers of compliance. The concentration of very long change saturated fatty acids will be analyzed in capillary blood micro-samples by HS-GC-MS in the 30% of the volunteers at baseline and after 6 months of intervention as biomarkers of compliance. Adherence levels will be considered in the statistical analysis.
* To determine the circulating levels of vascular risk factor, satiety hormones and inflammation parameters.

The investigators will evaluate the levels of adiponectin, adipsin, C-peptide, ghrelin, GIP, GLP-1, glucagon, insulin, leptin, PAI-1, resistin, and visfatin, interleukin 6 (IL -6), interleukin-10 (IL-10), and monocyte chemotactic protein 1 (MCP-1) by ELISA - Multiplex immunoassays. Moreover, TXA2 and PGI2 will be analysed in urine samples.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will be young adolescents, boys and girls, aged between 10 and 12 years who attend regular primary schools in Barcelona. The schools will assist with the participant recruitment through the classes and after that, a total of one-hundred students will be randomly included in each group. In all cases, participation will be voluntary and informed consent will be obtained prior to the study.

Exclusion Criteria:

The exclusion criteria will be history of allergy or intolerance to peanuts, any medical conditions or dietary restrictions that would affect peanut consumption, being able to understand Spanish or Catalan, and use of antibiotics in the month prior to the study.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the depression score in healthy young adolescents after a daily intake of peanuts. | Baseline and after 6 months
  To measure depression score, the CDI Childhood Depression Inventory test will be used.
Changes in the ability to concentrate, selective attention and processing speed in healthy young adolescents after a daily intake of peanuts. | Baseline and after 6 months
  To measure the ability to concentrate, selective attention and processing speed, the d2-R Attention Test (Revised) will be used.
Changes in assessment of interference and cognitive control in healthy young adolescents after a daily intake of peanuts. | Baseline and after 6 months
  To measure the assessment of interference and cognitive control, the Stroop test will be used.
Changes in processing speed, attention span and working memory in healthy young adolescents after a daily intake of peanuts. | Baseline and after 6 months
  To measure processing speed, attention span and working memory, the WISC-V Digits and Codes Subtest will be used.
Changes in attention and inductive reasoning in healthy young adolescents after a daily intake of peanuts. | Baseline and after 6 months
  To measure in attention and inductive reasoning, the Raven-2 test will be used.
Changes in Social cognition (emotion recognition and theory of mind) in healthy young adolescents after a daily intake of peanuts. | Baseline and after 6 months
  To measure Social cognition (emotion recognition and theory of mind), the NEPSY-II subtest will be used.
Changes in pro- and anti-inflammatory biomarkers after a daily intake of peanuts in healthy young adolescents. | Baseline and after 6 months
  Cytokines (pg/mL), Monocyte chemoattractant protein-1 (MCP-1) (pg/mL), interleukin (IL)-6 and 10 (pg/mL), (mg/dL) will be assayed by immunoenzymatic methods.
Changes in vascular biomarkers after a daily intake of peanuts in healthy young adolescents. | Baseline and after 6 months
  sVCAM-1 and sICAM-1 (ug/mL) will be assayed by immunoenzymatic methods.
Changes in adiposity molecules after a daily intake of peanuts in healthy young adolescents | Baseline and after 6 months
  Adiponectin and adipsin (ug/mL), leptin (pg/mL), ghrelin (pg/mL), visfatin (pg/dL), resistin (pg/mL), insulin (pg/mL), glucagon (pg/dL), peptid C (pg/mL) and, PAI-1 (pg/mL) will be assayed by immunoenzymatic methods.
Changes in body mass index after a daily intake of peanuts in healthy young adolescents | Baseline, 3 and after 6 months
  Body mass index (kg/m^2) are calculated after measure weight (kg) and height (meter).

SECONDARY OUTCOMES:
Changes in waist circumference after a daily intake of peanuts in healthy young adolescents | Baseline, 3 and after 6 months
  Change in waist circumference (cm) will be measured in triplicate
Changes in blood pressure after a daily intake of peanuts in healthy young adolescents | Baseline, 3 and after 6 months
  Systolic and diastolic blood pressure (mmHg) will be measured using an automatic blood pressure monitor in triplicate.
Changes in heart rate after a daily intake of peanuts in healthy young adolescents | Baseline, 3 and after 6 months
  Heart rate (bpm) is measured with an automatic monitor in triplicate.
Changes in lipidic profile after a daily intake of peanuts in healthy young adolescents | Baseline and after 6 months
  Total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides (mg/dL) will be measured using a portable Cardiocheck analyzer, through 40 µL of capillary and fasting blood.
Changes in blood glucose after a daily intake of peanuts in healthy young adolescents | Baseline and after 6 months
  Fasting blood glucose (mg/dL) will be measured using a portable Cardiocheck analyzer
Changes in nutrients and energy intake after regular peanut in healthy young adolescents | Baseline and after 6 months
  Dietary changes will be evaluated using a 151-item semi-quantitative food frequency questionnaire (Fernández-Ballart et al., 2010).
Changes in physical activity after regular peanut in healthy young adolescents | Baseline and after 6 months
  To study the association between changes in physical activity and changes in adiposity parameters . Actigraph wGT3X-BT accelerometers that allow the registration of the amount and intensity of physical activity will be used during 7 days per evaluation time-point. To complete this information a diary with questions about the type of physical activity performed during the 7 days will be collected. A validated questionnaire will be also used to assess physical activity habits (Barbosa et al., 2007).
Changes in sleep quality after regular peanut in healthy young adolescents | Baseline and after 6 months
  To study the association between changes in sleep quality and changes in adiposity parameters . Actigraph wGT3X-BT accelerometers that allow the registration of the amount and intensity of physical activity will be used during 7 days per evaluation time-point. To complete this information a diary with questions about the type of physical activity performed during the 7 days will be collected.
Pubertal changes in healthy young adolescents after a daily intake of peanuts. | Baseline and after 6 months
  To measure pubertal changes, the Tanner's Pubertal scale self-assessment questionnaire will be used.
Changes in the gut microbiota after a daily intake of peanuts in fecal samples of healthy young adolescents. | Baseline and after 6 months
  Fecal samples will be collected by the volunteers using a system for easy self-collection and stabilization of microbial DNA for gut microbiome profiling (OMNIgene - GUT). The genomic DNA will be extracted from fecal samples using the DNeasy PowerSoil Kit. Then, the 16s metagenomic analysis will be performed.
Changes in the short-chain fatty acids after a daily intake of peanuts in biological samples of healthy young adolescents. | Baseline and after 6 months
  After acidifying the fecal samples with formic acid, a quantification of short-chain fatty acids will be performed using gas chromatography by direct injection according to previously described methodology (Zhao et al., 2006).
Changes in the polyphenols and their metabolites after a daily intake of peanuts in biological samples of healthy young adolescents. | Baseline and after 6 months
  Identification and quantification of polyphenols will be determined using a high performance liquid chromatography-high resolution mass spectrometry (HPLC-HRMS) (Laveriano-Santos et al., 2022) and by ultra high-performance liquid chromatography coupled with triple quadrupole mass spectrometry (UHPLC-QqQ-MS/MS) (Martínez-Huélamo et al., 2015) methods.
Changes in percentage of body fat in healthy young adolescents after a daily intake of peanuts. | Baseline, 3 and after 6 months
  Total adiposity are measured by bioelectrical impedance (body fat %, muscle mass %, visceral fat (kg), fat mass index (kg/m^2), lean mass index (kg/m^2)).

CONTACTS AND LOCATIONS:
Locations (1):
- IDIBAPS, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
The dataset analyzed during the current study is not publicly available due to national data regulations and for ethical reasons, e.g. we do not have the explicit written consent of the study volunteers to make their deidentiﬁed data available at the end of the study. However, data described in the manuscript, codebook, and analytic codes will be made available upon request by contacting the PI and Co-PI (peanuty2023@gmail.com). The request will be passed to all the members of the study for deliberation.